CLINICAL TRIAL: NCT05390567
Title: Project CONTINUITY: Promoting Evidence-Based Cancer Screening Among Underserved Women
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202200613; OCR41931 (Other: UF OnCore)
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer Screening Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of Care in-clinic Pap-Test: Participant cervical cancer screening method of choice: Standard of Care Pap-Test
  Interventions: Behavioral: Survey: Participant cancer history and cervical cancer prevention/screening knowledge; Behavioral: Participant Choice of Standard of Care in-clinic Pap-test
- HPV Self-Test: Participant cervical cancer screening method of choice: HPV Self-Test
  Interventions: Behavioral: Participant Choice of HPV Self-Test; Behavioral: Survey: Participant cancer history and cervical cancer prevention/screening knowledge

INTERVENTIONS:
Behavioral: Participant Choice of HPV Self-Test — Opportunity for participants to complete the HPV self-test in a non-clinical setting to be returned via a mailer or courier servie.
  Groups: HPV Self-Test
Behavioral: Survey: Participant cancer history and cervical cancer prevention/screening knowledge — Asking women to respond to questions about their cancer history and knowledge of cervical cancer prevention and screening.
Behavioral: Participant Choice of Standard of Care in-clinic Pap-test — Participant choice of cervical cancer screening method with either a SOC in-clinic pap test or HPV self-test
  Groups: Standard of Care in-clinic Pap-Test

SUMMARY:
Project CONTINUITY (Connecting You to Care in the Community) was developed to increase adherence to cervical cancer screening regimens from initial screening to needed follow-up care by (1) providing personalized approaches to improve adherence through the combined use of patient choice for the initial screening method (Pap/HPV co-testing vs. HPV self-test collection), community clinical navigators and community health workers (CHWs), customized messages and support for patient portal access for test results and (2) implementing strategies to address social determinants of health (SDoH) that may influence an individual's ability to adhere to the screening regimen, with an initial focus on removing transportation barriers through the use of a mobile outreach clinics (MOC).

DETAILED DESCRIPTION:
The purpose of this pilot project is to gather information about the extent to which women residing in high SEV neighborhoods who choose HPV self-sampling relative to in-clinic Pap/HPV testing adhere to the cancer screening continuum steps, for which they are eligible. The women will self-select into HPV self-sampling versus in-clinic Pap/HPV testing combined with follow-up telephone calls and text messages from community clinical navigators and CHWs.

The research components of this study involve: 1) offering women the opportunity to complete the HPV self-test in a non-clinical setting to be returned via a mailer or handed to the community clinical navigator or CHW and 2) asking women to respond to questions about their cancer history and knowledge of cervical cancer prevention and screening. All other components of this study are part of clinical care. All other planned activities align with clinically based recommendations and guidelines (e.g., follow-up for colposcopy for + Paps)

ELIGIBILITY:
Inclusion Criteria:

1. Using the American Cancer Society (ACS) screening recommendations, adults 25 to 65 will be eligible.
2. Assigned sex at birth is female
3. No previous history of cervical cancer
4. No previous history of a hysterectomy
5. Not currently pregnant (self-report)
6. Not currently menstruating*
7. Have not used any vaginal products (e.g., oil-based lubricants, antifungal, and douches) in prior 2 days*. Use of vaginal contraceptives, condoms and water-based lubricants are allowed.
8. Have not given birth in the prior 12 weeks*
9. Self-report they have not undergone cancer screening in the past 4 years or more OR report being past due according to provider recommended screening schedule.
10. Self-report of using the MOC in the past, no current usual source of care OR usual source of care is a non-UFH provider and/or cervical cancer screening is not accessible through that provider
11. Reside in census tracts where the Mobile Outreach Clinic travels.
12. Have a mobile phone or access to a mobile phone that can be used to receive messages or a valid email address.

Exclusion Criteria:

* For patients who are excluded for criterion 6, 7, and 8, the outreach team (community clinical navigator and CHW) will ask the participant if they can be re-contacted for potential future study eligibility assessment. If the participant agrees, the navigator or CHW will collect contact information to re-contact the participant at a later (pre-determined) date up to 20 weeks later for eligibility screening.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned sex at birth is female
Study Population: Adults age 25 to 65 years old whose assigned sex at birth is female.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to steps in the cervical cancer screening continuum | 6 months
  For the HPV self-testing group,
  1. HPV test returned (Yes or No)
  2. Results obtained (Yes or No)
  3. Follow-up Pap test completed among those who tested positive for HPV (Yes or No)
  4. Follow-up colposcopy completed among those who had positive Pap test (Yes or No) For the in-clinic testing group,
  1. In-clinic Pap test completed (Yes or No) 2. Results Obtained (Yes or No) 3. Follow-up colposcopy completed among those who had positive Pap test (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi A Salloum, PhD, Principal Investigator — Division Director, Department of Health Outcomes and Biomedical Informatics, University of Florida; Associate Director, Office of Community Outreach and Engagement, UFHealth Cancer Center
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No